CLINICAL TRIAL: NCT01884220
Title: A Historical Chart Review and Longitudinal Follow-Up of Identified Patients With Wolman Disease or Cholesteryl Ester Storage Disease, Lysosomal Acid Lipase Deficiency
Brief Title: Wolman/CESD Natural History Chart Review and Longitudinal Follow-Up
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Center for Advancing Translational Sciences (NCATS) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: LDN6706; U54NS065768 (NIH)
Record Dates: First submitted 2013-03-13; First posted 2013-06-21 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Wolman Disease; Cholesterol Ester Storage Disease; Acid Cholesteryl Ester Hydrolase Deficiency, Type 2
Keywords: Wolman Disease; Cholesteryl Ester Storage Disease; Enzyme deficiency; Natural History; Medical Records Review
MeSH Terms: conditions — Wolman Disease; Cholesterol Ester Storage Disease

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: None Retained — No biospecimens will be collected specifically for this study. However, participants are encouraged to send left over biopsy material to the study site for analysis at a later date.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Disease: Patients with Wolman disease (WD), Cholesteryl Ester Storage Disease (CESD), or Lysosomal acid lipase (LAL) deficiency.
  Interventions: Other: There are no interventions in this study.

INTERVENTIONS:
Other: There are no interventions in this study.

SUMMARY:
The purpose of this study are: to characterize and understand the natural history of disease progression in WD and CESD, and to provide historical controls for WD and CESD for developing clinical treatment trials. The hypothesis is that the variability and clinical progression in WD and CESD is large and represents a continuum of severities from a lethal infantile to near normal adults with only "fatty livers".

DETAILED DESCRIPTION:
This is a single institution historical cohort study of patients with Wolman (WD) or Cholesteryl Ester Storage Disease (CESD). Retrospective data will be collected and abstracted from the medical records of both living and deceased patients. Additionally prospective data from living patients will be collected and abstracted annually until the end of the study. Literature sources will be used as secondary source data and will be screened to minimize/eliminate duplicative reports.

ELIGIBILITY:
Inclusion Criteria:

* male or female of any age;
* a clinical diagnosis of WD or CESD as defined by:

  * documented LAL enzyme deficiency OR
  * LAL gene mutations OR
  * a clinical course and tissue biopsy consistent with CESD or WD;
* written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited initially from the PIs patient population. Other physicians may refer their patients to this study for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2010-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Organ Measurements using Ultrasound Imaging | Baseline, Year 1, Year 2, Year 3, Year 4
  Measurement of the effect over time of LAL deficiency on the liver, spleen, intestines, lungs and adrenals will be performed using ultrasound imaging. Measurement using ultrasound imaging will only be completed if clinically indicated during clinical-care patient visits.

SECONDARY OUTCOMES:
Change in Organ Measurements using X-Ray Imaging | Baseline, Year 1, Year 2, Year 3, Year 4
  Measurement of the effect over time of LAL deficiency on the liver, spleen, intestines, lungs and adrenals will be performed using X-rays. Measurement using X-ray imaging will only be completed if clinically indicated during clinical-care patient visits.
Change in Organ Measurements using Computerized Tomography | Baseline, Year 1, Year 2, Year 3, Year 4
  Measurement of the effect over time of LAL deficiency on the liver, spleen, intestines, lungs and adrenals will be performed using Computerized Tomography. Measurement using Computerized Tomography imaging will only be completed if clinically indicated during clinical-care patient visits.
Change in Organ Measurements using Magnetic Resonance Imaging | Baseline, Year 1, Year 2, Year 3, Year 4
  Measurement of the effect over time of LAL deficiency on the liver, spleen, intestines, lungs and adrenals will be performed using Magnetic Resonance Imaging. Measurement using Magnetic Resonance Imaging will only be completed if clinically indicated during clinical-care patient visits.
Change in Liver Function using Standardized Laboratory Liver Function Assessment | Baseline, Year 1, Year 2, Year 3, Year 4
  Measurement of the effect over time of LAL deficiency on the liver will be performed using standardized laboratory liver function assessments during clinical-care visits.
Change in Pulmonary Function using Standardized Pulmonary Function Assessment | Baseline, Year 1, Year 2, Year 3, Year 4
  Measurement of the effect over time of LAL deficiency on the lungs will be performed using standardized pulmonary function assessment during clinical care visits. Measurement using standardized pulmonary function assessment will only be completed if clinically indicated during clinical-care patient visits.
Change in Subjects's Overall Health Status using Clinical Exam | Baseline, Year 1, Year 2, Year 3, Year 4
  Measurement of the effect over time of LAL deficiency on the subject's physical health status will be performed using clinical physical exams during clinical-care visits.
Change in the Subject's Overall Health Status using Verbal Report | Baseline, Year 1, Year 2, Year 3, Year 4
  Measurement of the effect over time of LAL deficiency on the subject's overall health status will be performed using patient's or parents' verbal report during clinical-care visits.

CONTACTS AND LOCATIONS:
Overall Officials: Gregory A Grabowski, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States